CLINICAL TRIAL: NCT00245440
Title: Influence of Oral Telithromycin vs. Azithromycin on the Endogenous Microflora in Adults With Acute Sinusitis
Brief Title: Study to Measure the Impact of Antibiotics on Bacterial Flora in Adults With Acute Sinusitis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor Terminated
Sponsor: CPL Associates (Other)
Collaborators: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HMR3647A-6045
Record Dates: First submitted 2005-10-26; First posted 2005-10-28 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Maxillary Sinusitis
Keywords: S.pneumonia; sinusitis; ams; azithromycin
MeSH Terms: conditions — Maxillary Sinusitis; Sinusitis; Focal Facial Dermal Dysplasias | interventions — Azithromycin; telithromycin

ARMS (2):
- 1 (Active Comparator): Subjects assigned Azithromycin
  Interventions: Drug: Azithromycin
- 2 (Active Comparator): Subjects assigned Telithromycin
  Interventions: Drug: Telithromycin

INTERVENTIONS:
Drug: Azithromycin — 250 mg tablets; 2 tablets once daily (500 mg) for 3 days
  Arms: 1
Drug: Telithromycin — 400 mg tablets; 2 tablets once daily (800 mg) for 5 days
  Arms: 2

SUMMARY:
The purpose of this study is to measure the speed of microbial eradication due to azithromycin or telithromycin in acute maxillary sinusitis (AMS).

DETAILED DESCRIPTION:
The objectives of this study are:

* To assess the impact of therapy with telithromycin vs. azithromycin on the oral microflora in patients with acute maxillary sinusitis at day 42 and to compare the duration of colonization with resistant oropharyngeal flora in patients treated with azithromycin vs. telithromycin.
* To also compare the two treatment groups for rate of reinfection within 6 weeks and the susceptibility pattern of the organisms appearing during the reinfection and differences in development of resistance and the associated changes in symptom responses.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, either males or non-pregnant females, aged 18 to 75 years of age with clinical findings of acute maxillary sinusitis (AMS), who are amenable to serial sampling of the nasopharynx and oropharynx.
* Patients are required to have specimens of nasal and nasopharyngeal drainage collected for microbiological documentation within 24 hours prior to enrollment. All patients must produce sinus fluid drainage.
* All patients will produce nasal or nasopharyngeal discharge sufficient for baseline culture.
* Female patients of child bearing potential must agree to use an accepted method of contraception (i.e., oral or implanted contraceptive with a barrier method, spermicide and barrier methods, or intrauterine device [IUD]). The patient must agree to continue with the same method throughout the study.

Exclusion Criteria:

* Patients with a history of recurrent sinusitis defined as more than three episodes of sinusitis which required antibiotic therapy in the preceding 12 months
* Patients with a history of chronic sinusitis defined as symptoms lasting greater than 28 days
* Patients with nosocomial acquired sinusitis (e.g., hospitalization or non-ambulatory institutional confinement including nursing homes within 2 weeks)
* Patients with a need for immediate surgery for maxillary sinusitis or previous sinus surgery within the past 6 months or sinus lavage within the past 7 days
* Patients who are long-term (> 4 weeks) users of nasal decongestants (e.g. oxymetazoline 0.05%)
* Patients with a known or suspected hypersensitivity to, or a known or suspected serious adverse reaction to, any macrolide antibiotic
* Impaired hepatic or renal function (creatinine clearance [CCL] <20 ml/min)
* Severe respiratory tract infections requiring hospitalization and parenteral antibiotic therapy.
* Requirement for a concomitant antimicrobial agent other than topical, antiviral or antifungal agents.
* Treatment with any macrolide, azalide, or ketolide antimicrobial within the 30 days prior to entry into the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2005-12; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Bacterial resistance or selection | 42 days

SECONDARY OUTCOMES:
Bacteriologic outcome | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Jerome J Schentag, Pharm.D., Principal Investigator — State University of NY at Buffalo; Joseph Paladino, Pharm.D., Study Director — State University of NY at Buffalo
Locations (1):
- Southeastern Researchs Associates,Inc., Taylors, South Carolina, United States

REFERENCES:
- See also: Related Info — http://www.cplassociates.com